CLINICAL TRIAL: NCT04933552
Title: Post-Authorization Safety Study for Assessment of Pregnancy Outcomes in Patients Treated With Mayzent (Siponimod): An OTIS Observational Pregnancy Surveillance Study
Brief Title: Post-Authorization Safety Study for Assessment of Pregnancy Outcomes in Patients Treated With Mayzent
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312A2403
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; PASS; Post-Authorization Safety Study; Mayzent; Siponimod; Pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — siponimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Siponimod-Exposed: Pregnant women with MS exposed to siponimod during pregnancy
  Interventions: Other: Siponimod
- Disease-Matched Comparison: Pregnant women with MS not exposed to siponimod during pregnancy
- Healthy Comparison: Pregnant women who are neither diagnosed with MS nor with any other autoimmune disease, and not exposed to siponimod or any known teratogenic agent during pregnancy

INTERVENTIONS:
Other: Siponimod — Prospective observational cohort study. There is no treatment allocation. Patients administered siponimod, that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Mayzent
  Groups: Siponimod-Exposed

SUMMARY:
This study will utilize a prospective, observational, exposure cohort design to examine pregnancy and infant outcomes in women and infants who are exposed to siponimod during pregnancy to treat MS.

DETAILED DESCRIPTION:
The prevalence of each outcome in women exposed to siponimod and their infants will be compared to those observed in two unexposed comparator groups: a disease-matched comparison group of women who have not used siponimod during pregnancy but have been diagnosed with MS (disease-matched unexposed comparison group), and a comparison group of healthy women who do not have diagnosis of MS, have not had exposure to a known human teratogen, and have not taken siponimod in pregnancy (healthy comparison group). Pregnant women exposed to siponimod who do not meet the prospective cohort criteria will also be followed as part of an exposure series. All participants will be recruited via voluntary participant registration following informed consent by the pregnant woman for her participation. Participants may withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the criteria listed under the respective cohorts to enroll in that particular cohort of the registry:

Cohort 1: Siponimod-Exposed Cohort

1. Pregnant women
2. Diagnosed with MS, with the indication validated by medical records when possible
3. Exposure to siponimod for the treatment of MS, for any number of days, at any dose, and at any time from the 4th day post the first day of LMP prior to conception up to and including the end of pregnancy
4. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants, and the Ages and Stages Questionnaire (ASQ) in live born children

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1)

1. Pregnant women
2. Diagnosed with MS, with the indication validated by medical records when possible
3. May or may not have taken another medication for MS in the current pregnancy
4. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants, and the ASQ in live born children

Cohort 3: Healthy Comparison Cohort (Comparison Group 2):

1. Pregnant women
2. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants, and the ASQ in live born children

Exclusion Criteria:

Women meeting any of the following criteria will be excluded from the cohort study:

Cohort 1: Siponimod-Exposed Cohort

1. Women who have enrolled in the siponimod cohort study with a previous pregnancy
2. Women who have used siponimod for an indication other than a currently approved indication
3. Women with exposure to any of the following medications within 5 half-lives prior to conception:

   * Cladribine (Mavenclad)
   * Based on the US label, animal studies indicate that there is positive evidence of teratogenicity for Cladribine
   * All other S1P modulators including fingolimod (Gilenya), ozanimod, etc.
   * S1P modulatros are in the same class of drug as siponimod
   * Teriflunomide (Aubagio)
   * The teratogenicity of teriflunomide is unknown and currently under investigation
   * Other anti-CD20 monoclonal antibody: same class as Kesimpta
   * New medications (marketed after 2020) indicated for the treatment of MS will be evaluated for inclusion/exclusion criteria as the study progresses.
4. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
5. Results of a diagnostic test are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1):

1. Exposure to siponimod any time from the 4th day post the first day of LMP prior to conception up to and including end of pregnancy
2. Women with exposure to any of the following medications within 5 half-lives of conception:

   * Cladribine (Mavenclad)
   * S1P modulators
   * Teriflunomide (Aubagio)
   * Anti CD-20 monoclonal antibody New medications (marketed after 2020) indicated for the treatment of MS will be evaluated for inclusion/exclusion criteria as the study progresses.
3. Women who have enrolled in the siponimod cohort or OMB157G2403 Kesimpta cohort with a previous pregnancy
4. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
5. Results of a diagnostic test are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Cohort 3: Healthy Comparison Cohort (Comparison Group 2):

1. Exposure to Kesimpta 166 days before or to siponimod any time from the 4th day post first day of LMP prior to conception to and including end of pregnancy
2. Women who have a diagnosis of a MS or a siponimod approved indication
3. Women who have a current diagnosis of any autoimmune disease
4. Women who have first contact with the project after prenatal diagnosis of any major structural defect
5. Women who have enrolled in the siponimod cohort or Kesimpta cohort study with a previous pregnancy
6. Women treated with Mayzent or Kesimpta for non-MS indication
7. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
8. Results of a diagnostic test are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.
9. Women exposed to a known human teratogen during pregnancy as confirmed by the OTIS Research Center

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study population includes pregnant women.
Study Population: The study population includes pregnant women who reside in the US or Canada.
Sampling Method: Non-Probability Sample
Enrollment: 867 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of major structural defects | Up to 10,5 years
  A major structural defect is defined as a defect that has either cosmetic or functional significance to the child (e.g., a cleft lip).

SECONDARY OUTCOMES:
Number of spontaneous abortion/miscarriage | Up to 10,5 years
  Spontaneous abortion/miscarriage is defined as non-deliberate fetal death which occurs prior to less than 20.0 weeks post-LMP.
Number of stillbirth | Up to 10,5 years
  stillbirth is defined as non-deliberate fetal death anytime in gestation at or after 20 weeks post-LMP.
Number of elective termination | Up to 10,5 years
  elective termination/abortion is defined as deliberate termination of pregnancy at any time in gestation. Reasons for elective abortions are captured and are classified as due to medical reasons or social reasons.
Number of premature delivery | Up to 10,5 years
  premature delivery is defined as live birth prior to 37.0 weeks gestation as counted from LMP (or calculated from first-trimester ultrasound-derived due date if last menstrual period uncertain or more than 1 week discrepant). Elective caesarian deliveries or inductions prior to 37.0 completed weeks will be considered separately.
Number of preeclampsia / eclampsia | Up to 1 10,5 years
  preeclampsia or eclampsia reported by maternal interview with confirmation in medical record or report by medical record only is captured.
  Preeclampsia is defined as a new onset of hypertension and proteinuria during pregnancy or postpartum. Eclampsia is the new onset of seizures or coma in a pregnant woman with preeclampsia. These seizures are not related to an existing brain condition.
Pattern of 3 or more minor structural defects | Up to 10,5 years
  A minor structural defect is defined as a defect which has neither cosmetic nor functional significance to the child (e.g., complete 2,3 syndactyly of the toes). Minor structural defects will be identified only through the study dysmorphology examination for live born infants using the study-specific checklist.
Small for gestational age | Up to 10,5 years
  small for gestational age is defined as birth size (weight, length or head circumference) less than or equal to the 10th centile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants (CDC, 2000; Olsen et al., 2010).
Postnatal growth small for age at approximately one year of age | Up to 10,5 years
  postnatal growth deficiency is defined as postnatal size (weight, length or head circumference) less than or equal to the 10th centile for sex and age using National Center for Health Statistics (NCHS) pediatric growth curves, and adjusted postnatal age for premature infants if the postnatal measurement is obtained at less than one year of age (CDC, 2000).
Developmental performance at approximately one year of age | Up to 10,5 years
  Screening of Developmental Milestones: one or more domains scored as abnormal on the Ages and Stages Questionnaire completed by the mother when the infant is approximately one year of age will define achievement of developmental milestones.
Serious or opportunistic infections in the first year of life | Up to 10,5 years
  serious or opportunistic infections are defined as any one or more diagnoses of tuberculosis, x-ray proven pneumonia, neonatal sepsis, meningitis, bacteremia, invasive fungal infection, pneumocysitis, septic arthritis, osteomyelitis, abcess (deep tissue), and infections requiring hospitalization identified in live born infants up to one year of age.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MotherToBaby Pregnancy Studies are observational studies coordinated at the University of California San Diego. Our studies are currently enrolling pregnant women in a study examining the use of medications to treat multiple sclerosis during pregnancy. — https://mothertobaby.org/ongoing-study/mayzent-siponimod/